CLINICAL TRIAL: NCT01772030
Title: Mechanisms and Patterns of Atrial Fibrillation Recurrence After Cryoballoon Ablation
Brief Title: Atrial Fibrillation Recurrence After Cryoballoon Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Sandeep Jain, Associate Professor of Medicine, Cardiac Electrophysiology, University of Pittsburgh, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO12060524
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Cryoballoon Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recurrent Atrial Fibrillation (Other)
  Interventions: Other: Use of the Achieve catheter followed by ICE-guided mapping catheter

INTERVENTIONS:
Other: Use of the Achieve catheter followed by ICE-guided mapping catheter

SUMMARY:
The purpose of the study is to evaluate the mechanisms of recurrent atrial fibrillation after cryoballoon ablation using the Arctic Front Ablation System. For those with pulmonary vein reconnection, specific sites of reconnection will be evaluated with left atrial intracardiac echo (ICE) guidance. The Achieve mapping catheter will be evaluated head-to-head with our current method of ICE-guided recordings from a conventional mapping catheter with high output pulmonary venous pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing re-do catheter ablation procedure after index procedure with cryoballoon ablation
* At least 18 years old
* Able to read and understand informed consent

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Presence or absence of pulmonary vein isolation or reconnection | During repeat cryoballoon ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep K Jain, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania